CLINICAL TRIAL: NCT03999983
Title: Vertebral Artery Origin Treatment Via Endovascular Techniques Registry (VOTER)
Acronym: VOTER
Status: Recruiting | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Randall C. Edgell, MD, FSVIN, Professor, Department of Neurology, St. Louis University
Other Study IDs: 29760
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Vertebral Artery Stenosis
MeSH Terms: conditions — Vertebrobasilar Insufficiency | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational Prospective Registry — This is a prospective registry looking at patients admitted for stroke with evidence of Vertebral Artery Origin Stenosis. Patients clinical outcomes will be collected at 30 days and 1-year post-treatment and angiographic outcomes at 1-year post-treatment
  Other Names: Observational

SUMMARY:
A retrospective and prospective registry of patients admitted for stroke and evidence of Vertebral Artery Origin Stenosis (VAOS).

DETAILED DESCRIPTION:
A retrospective registry of stenting plus medical management for the prevention of recurrent stroke in patients with symptomatic Vertebral Artery origin Stenosis (VAOS). This study is collecting information on clinical outcomes up to 18 months post-treatment.

On January 6, 2025, VOTER was changed from prospective to retrospective.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 90 years of age
2. Patient has experienced a posterior circulation ischemic event
3. Patient has angiographically confirmed bilateral vertebral artery origin disease (Hypoplasia, occlusion, or stenosis).
4. Patient has >50% stenosis on the side being targeted for therapy

Exclusion Criteria:

1. Pregnant women
2. Contrast Indication to the use of anti-platelet drugs
3. There is tandem vertebral or basilar artery stenosis
4. The serum creatinin is >2.5
5. Baseline modified Rankin score is >3
6. < 5 years life expectancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for stroke and evidence of Vertebral Artery Origin Stenosis (VAOS).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of recurrent stroke or death | 1 Year post-treatment
  Recurrent stroke of any type or death from any cause

SECONDARY OUTCOMES:
Incidence of Restenosis | 1 Year post-treatment
  Restenosis in VAOS patients treated with drug-eluting stents.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Edgell, MD, Principal Investigator — St. Louis University
Locations (10):
- United States (10):
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - University of Southern Florida, Tampa, Florida
  - Northwestern Medicine Regional Medical Group, Winfield, Illinois
  - University of Iowa, Iowa City, Iowa
  - SSM DePaul Hospital, Bridgeton, Missouri
  - Saint Louis University, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Mercy Health Neuroscience Institute, Toledo, Ohio
  - Semmes Murphey Clinic, Memphis, Tennessee
  - Texas Tech University Health Science Center of El Paso, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Undecided